CLINICAL TRIAL: NCT05429957
Title: Effects of Muscle Energy Technique Versus Aerobic Exercises on Pain and Disability in Patients With Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0516
Record Dates: First submitted 2022-06-20; First posted 2022-06-23 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Pain; Chronic Pain
Keywords: Pelvic Pain; Female; Exercise
MeSH Terms: conditions — Pelvic Pain; Chronic Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental): Muscle Energy Technique of Iliopsoas, Piriformis, Quadratus Lumborum and Erector Spinae muscle
  Interventions: Other: Muscle Energy Technique
- Aerobic Exercises (Experimental): aerobic exercises (walking on the treadmill)
  Interventions: Other: Aerobic Exercises

INTERVENTIONS:
Other: Muscle Energy Technique — Muscle energy technique (Post Isometric relaxation) three times per week for 8 weeks.
  * MET of the Iliopsoas
  * MET of Piriformis muscle
  * MET of Quadratus Lumborum muscle
  * MET of Erector Spinae muscle
  Arms: Muscle Energy Technique
Other: Aerobic Exercises — Aerobic exercise (treadmill walking) three times per week for 8 weeks
  * Warm-up phase: in which each patient alternately steps their legs forward, backward, and sideways in each direction for 5 min
  * Active phase: Treadmill speed was 3km/hour for 5 weeks and progress to 4km/hour after 5 weeks for 20 min.
  * Cool down phase: During a cool down period take a deep breath with both arms overhead and exhale while bringing the arms down, shaking out the legs and arms for 5 min.
  Arms: Aerobic Exercises

SUMMARY:
The aim of study is to find out the effects of muscle energy technique versus aerobic exercises on pain and disability in patients with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* women with chronic pelvic pain of >6 months' duration and the cause of their pain is unknown
* CPP was located within the true pelvis (between and below the anterior iliac crests)
* Average score of at least 4 out of 10 (0-10) on a numeric rating scale
* moderate to severe pain on pelvic pain impact questionnaire

Exclusion Criteria:

* History of cancer
* Pregnancy at the time of inclusion
* Known pelvic pathology (eg, endometriosis, ovarian cyst, fibroid >3cm)
* Intraabdominal and pelvic surgery within the last six months
* chronic or recurrent gastro-intestinal disease including irritable bowel syndrome
* Received any physiotherapy treatment within the previous month

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pelvic pain is more common in female
Enrollment: 40 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Pelvic pain impact questionnaire | 8th week
  The Pelvic Pain Impact Questionnaire evaluates the pelvic pain impact on life. It has patient generated language, is easily managed and scored, has psychometric properties and it is appropriate for clinical settings and research across primary, secondary and tertiary care. The ten-item questionnaire consist of 8 Likert questions and 2 additional, non-scored questions
Numerical Pain Rating Scale | 8th week
  The Numerical Pain Rating Scale (NPRS) is a particular measure in which people rate their pain on an 11-point numerical scale. The scale is comprised of 0 (no pain at all) to 10, 0 show no pain at all and 10 indicate worst imaginable pain

SECONDARY OUTCOMES:
Pain disability index | 8th week
  The Pain Disability Index is a seven-item survey to investigate functional disability. Every question utilizes an ordinal scale going from 0 to 10, 0 indicates no disability and 10 means worst disability. Scores can be added to represent a combined score of worldwide disability ranging from 0 to 70 ,where higher scores indicate greater disability

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam, MS, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuentes-Marquez P, Cabrera-Martos I, Valenza MC. Physiotherapy interventions for patients with chronic pelvic pain: A systematic review of the literature. Physiother Theory Pract. 2019 Dec;35(12):1131-1138. doi: 10.1080/09593985.2018.1472687. Epub 2018 May 14. PMID 29757068
- [Background] Chong OT, Critchley HO, Williams LJ, Haraldsdottir E, Horne AW, Fallon M. The impact of meridian balance method electro-acupuncture treatment on chronic pelvic pain in women: a three-armed randomised controlled feasibility study using a mixed-methods approach. Br J Pain. 2018 Nov;12(4):238-249. doi: 10.1177/2049463718776044. Epub 2018 May 14. PMID 30349698
- [Background] Horne AW, Vincent K, Hewitt CA, Middleton LJ, Koscielniak M, Szubert W, Doust AM, Daniels JP; GaPP2 collaborative. Gabapentin for chronic pelvic pain in women (GaPP2): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2020 Sep 26;396(10255):909-917. doi: 10.1016/S0140-6736(20)31693-7. PMID 32979978
- [Background] Ghai V, Subramanian V, Jan H, Pergialiotis V, Thakar R, Doumouchtsis SK; CHORUS: An International Collaboration for Harmonising Outcomes, Research, Standards in Urogynaecology, Women's Health. A systematic review on reported outcomes and outcome measures in female idiopathic chronic pelvic pain for the development of a core outcome set. BJOG. 2021 Mar;128(4):628-634. doi: 10.1111/1471-0528.16412. Epub 2020 Sep 1. PMID 32654406
- [Background] Lamvu G, Carrillo J, Ouyang C, Rapkin A. Chronic Pelvic Pain in Women: A Review. JAMA. 2021 Jun 15;325(23):2381-2391. doi: 10.1001/jama.2021.2631. PMID 34128995
- [Background] Nygaard AS, Stedenfeldt M, Oian P, Haugstad GK. Characteristics of women with chronic pelvic pain referred to physiotherapy treatment after multidisciplinary assessment: a cross-sectional study. Scand J Pain. 2019 Apr 24;19(2):355-364. doi: 10.1515/sjpain-2018-0308. PMID 30703061